CLINICAL TRIAL: NCT06287606
Title: A Prospective, Randomized, Investigator-blinded, Parallel, Multi-center, Phase 3 Trial in Bowel Preparation for Colonoscopy
Brief Title: A Phase 3 Clinical Trials for Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTP0302
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Bowel Preparation
Keywords: bowel preparation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CTP0302-A (Experimental): 2 days split-dose
  Interventions: Drug: CTP0302-A
- CTP0302-B (Experimental): One day dose
  Interventions: Drug: CTP0302-B
- Conventional OST (Active Comparator): 2 days split-dose
  Interventions: Drug: Conventional OST

INTERVENTIONS:
Drug: CTP0302-A — Subjects randomized into group CTP0302-A will take a bowel preparation from the evening until the following morning.
  Other Names: Treatment Group A
  Arms: CTP0302-A
Drug: CTP0302-B — Subjects randomized into group CTP0302-B will take a bowel preparation on the Colonoscopy day
  Other Names: Treatment Group B
  Arms: CTP0302-B
Drug: Conventional OST — Subjects randomized into group Conventional OST will take a bowel preparation from the evening until the following morning.
  Other Names: Control group
  Arms: Conventional OST

SUMMARY:
A prospective randomized study compared to the active control. Researchers compare colon cleansing in patients undergoing colonoscopy

DETAILED DESCRIPTION:
This is a prospective randomized study compared with active control arm. The investigators compare the colon cleansing in patients undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent.
* Male and female outpatients and inpatients aged: ≥19
* Patients BMI shoule be ≤ 30

Exclusion Criteria:

* Patients with past history of severe constipation (requiring repeated use of laxatives/enema or physical intervention before resolution), known or suspected ileus, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
* Patients with ongoing severe acute Inflammatory Bowel Disease.
* Patients who have had previous significant gastrointestinal surgeries, including colonic resection, subtotal colectomy, abdominoperineal resection, defunctioning colostomy.
* Pregnant women or pregnant women or pregnant women
* Severe heart disease (cardiac failure (NYHA class 3 and 4))
* Acute coronary artery disease within 24 weeks before screening (an unstable angina pectoris, acute myocardial infarction), clinically significant arrhythmia, hypertrophic obstruction Cardiomyopathy, valvular disease, aortic and peripheral vascular diseases.
* People who have hypersensitivity or allergies to clinical trial drug components.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Ratio of subjects With successful Bowel Cleansing | 1 day of scheduled colonoscopy
  The overall quality of bowel cleansing was assessed by a blinded central reader (an experienced and trained colonoscopist) using the segmental scores of the Harefield Cleansing Scale (HCS). A final HCS grading of A, B, C or D was derived. Grades A and B are classified as successful (i.e. all mucosa could be visualized) and C and D are classified as unsuccessful.

SECONDARY OUTCOMES:
Each segments ratio of subject with successful Bowel Cleansing | 1 day of scheduled colonoscopy
  Evaluate the HCS grade evaluation, polyp or adenoma detection rate, etc.

OTHER OUTCOMES:
Comparison of Acute gastropathy probability score | 1 day of scheduled colonoscopy
  According to 'The Manual of Gastric Mucosal Assessment', it's graded on a scale of 'Possible' to 'Very likely'.

CONTACTS AND LOCATIONS:
Overall Officials: Jaemyung Cha, MD. PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Taejoon Pharmaceutical Co., Ltd., Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SK, Jeon SR, Yang DH, Chun J, Cha JM. Efficacy and Safety of Bowel Cleansing with Mini S-Oral Sulfate Tablet versus the Conventional Oral Sulfate Tablet: A Prospective, Randomized, Investigator-Blinded, Multicenter, Noninferior, Phase 3 Trial. Gut Liver. 2025 Nov 27. doi: 10.5009/gnl250291. Online ahead of print. PMID 41306094